CLINICAL TRIAL: NCT02700308
Title: A Randomized, Multicenter, Open-label, Bayesian-based Phase II Study of the Feasibility of Kyphoplasty in the Local Treatment of Spine Metastases From Solid Tumors
Brief Title: A Study of Kyphoplasty and Vertebroplasty in the Treatment of Spine Metastases
Acronym: KYPHO-01
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DECISION OF THE SPONSOR AND THE COORDINATING INVESTIGATOR DUE TO RECRUITMENT DIFFICULTIES AND CHANGES IN INTERVENTIONAL RADIOLOGY PRACTICES
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET14000050
Record Dates: First submitted 2015-10-27; First posted 2016-03-07 (Estimated); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Solid Tumors; Spine Metastasis
Keywords: Solid tumors; Spine metastasis; Vertebroplasty; kyphoplasty; randomization
MeSH Terms: interventions — Kyphoplasty; Vertebroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional vertebroplasty (Active Comparator): Conventional vertebroplasty (device's trade at the discretion of the investigator)
  Interventions: Device: Conventional vertebroplasty
- Kyphoplasty (Experimental): Vertebroplasty with balloon placement and inflation prior to cement injection (device's trade at the discretion of the investigator)
  Interventions: Device: Kyphoplasty

INTERVENTIONS:
Device: Kyphoplasty — Placement and inflation of balloon prior to cement injection
  Other Names: Balloon kyphoplasty
  Arms: Kyphoplasty
Device: Conventional vertebroplasty — Conventional vertebroplasty
  Other Names: Vertebroplasty
  Arms: Conventional vertebroplasty

SUMMARY:
Conventional vertebroplasty is an effective option in the treatment of bone lesions (osteoporotic and neoplastic). It is indicated as an analgesic treatment and aims at reinforcing a compressed vertebrae or at risk of fracture.

The main adverse event related to vertebroplasty use is the cement leakages that might be responsible for significant clinical impairments.

Kyphoplasty is a recent alternative strategy of vertebroplasty, based on the insertion on balloon through the needle into the targeted vertebrae and then inflation of the balloon prior to cement injection into the space.

In an osteoporotic setting, kyphoplasty allow reducing the incidence of cement leakage.

To date, no data from randomized study are available in the population of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer other than malignant hemopathies, myeloma, brain tumors, germ-cell tumors and bone sarcomas;
* 2 metastatic sites or more;
* Spine metastasis between T1 and L5 with reduction of vertebrae of 20% at least;
* Indication of cementoplasty of 1 to 6 vertebrae defined by 1 of the following:
* Pain equal or greater than 4/10 at Visual Analogic Scale
* Unstable vertebrae (SINS score equal or greater than 7;
* Performance Status of the Eastern Cooperative Oncology Group : 0, 1 or 2

Exclusion Criteria:

* Contraindication to vertebroplasty, including contraindication to cement use;
* Patient already treated by vertebroplasty within the past 3 months (1 patient can not be allocated twice in this study);
* Previous focal treatment of the targeted vertebrae (vertebroplasty, percutaneous radiofrequency, embolization);
* Neurological deficit due to medullar or radicular compression;
* Participation to another clinical trial with an analgesic intent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Success rate for each strategy | 3 months after the procedure
  The success rate will be calculated with the proportion of patients without cement leakage

SECONDARY OUTCOMES:
Height of the targeted vertebrae | 3 months after the procedure
Height of the patient | 3 months after the procedure
Kyphotic angle | 3 months after the procedure
Analgesic properties of the strategies the day after the procedure | The day after the procedure
  Pain will be assessed using a Visual Analogic Scale
Analgesic properties of the strategies at 21 days | 21 days after the procedure
  Pain will be assessed using a Visual Analogic Scale
Analgesic properties of the strategies at the end of the study | 3 months after the procedure
  Pain will be assessed using a Visual Analogic Scale
Tolerance profile of the strategies | Through study completion
  Tolerance will be evaluated according to the National Cancer Institute - Common Terminology Criteria Adverse Event grading scale version 4
Type of cement leakage (vascular versus cortical localisation) | 3 months after the procedure
  Location will be described as vascular or cortical using the imaging assessments
Size of cement leakage | 3 months after the procedure
  Size will be described as significant or not significant as per investigator judgement
Symptoms associated with cement leakage | 3 months after the procedure
  Symptoms associated with cement leakage will be tolerance events that are stated by the investigator as related to a cement leakage
Quality of Life in both arms at Day 21 | 21 days after procedure
  Quality of Life will be assessed with the Dallas questionnaire for spinal pain
Quality of Life in both arms at the end oh study | 3 months after the procedure
  Quality of Life will be assessed with the Dallas questionnaire for spinal pain
Correlation between volume of cement injected and the level of pain relief using the Visual Analogic Scale | 3 months after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Amine BOUHAMAMA, MD, Principal Investigator — Centre Leon Berard
Locations (2):
- France (2):
  - Centre Léon Bérard, Lyon
  - Hopital Nord, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No